CLINICAL TRIAL: NCT04736576
Title: Prospective, Multicenter, Observational Study to Evaluate Patient-reported Outcome and Physical Activity Using Smartphone-based Application and Wearable Device in Japanese Patients With HR+/HER2- Advanced Breast Cancer Treated With Palbociclib Plus Endocrine Therapy or Endocrine Monotherapy
Brief Title: Study to Evaluate Patient Reported Outcome (PRO) and Physical Activity in Japanese Patients With HR+/HER2- Advanced Breast Cancer Treated With Palbociclib Plus Endocrine Therapy or Endocrine Monotherapy
Acronym: JBCRG-26
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Japan Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A5481126
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Prospective; Multicenter; Observational study; Japan; hormone receptor - positive/human epidermal growth factor 2 - negative (HR+/HER2-) advanced breast cancer; Palbociclib; European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-30 (items) (EORTC-QLQ-C30); Physical activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Palbociclib plus endocrine therapy
  Interventions: Device: Wearable device
- Group 2 (Other): Endocrine monotherapy
  Interventions: Device: Wearable device

INTERVENTIONS:
Device: Wearable device — As a low-interventional procedure, enrolled patients will be provided with wearable device and requested to wear the device at all-times, except of while bathing and sleeping, for 6 cycles (24 weeks).

SUMMARY:
The study is a prospective, multicenter, observational study to evaluate PRO and physical activity using smartphone-based application and wearable device in Japanese patients with HR+/HER2- advanced breast cancer (ABC).

Patients will be enrolled into either palbociclib plus endocrine therapy group (Group 1) or endocrine monotherapy group (Group 2) based on the discretion of the treating physician under routine clinical practice. Total target number of patients is approximately one-hundred in this study (About 50 patients in each group).

Enrolled patients will download a smartphone-based application for electronic PRO (ePRO), be provided access to and trained on the use of the application to complete baseline, weekly, and cycle-based assessments for 6 cycles (24 weeks). In addition, enrolled patients will be provided with wearable device and requested to wear the device at all-times, except of while bathing and sleeping, for 6 cycles (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥ 20 years of age)
2. Diagnosis of adenocarcinoma of the breast with evidence of metastatic disease or advanced disease not amenable to resection or radiation therapy with curative intent.
3. Documented evidence of HR+/HER2- tumor based on the patient's surgical specimen or most recent tumor biopsy.
4. Initiating first or second line treatment at study entry with one of the following therapies:

   palbociclib plus endocrine therapy or endocrine monotherapy
5. Eastern Cooperative Oncology Group (ECOG) performance status = 0~1.
6. Owns or has regular access to an Apple iPhone or Android phone.
7. Willing and able to complete collection of data via smartphone-based application.
8. Willing and able to wear the wearable device for approximately 6 months.
9. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
10. Able to read and understand Japanese

Exclusion Criteria:

1. The patient is participating in any interventional clinical trial that includes investigational or marketed products. Patients participating in other investigator-initiated research or non-interventional studies can be included as long as their standard of care is not altered by the study.
2. The patient is on active treatment for other malignancies other than ABC.
3. The patient's life style is fluctuating in weekly-basis (eg, shift-time worker), which may have high impact on physical activity assessment based to investigator's discretion

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 99 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Hiroko Bando, Principal Investigator — Dept of Breast, Thyroid and Endocrine Surgery, University of Tsukuba Hospital
Locations (20):
- Japan (20):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Sunagawa City Medical Center, Sunagawa, Hokkaido
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Sakai City Medical Center, Sakai, Osaka
  - Saitama Cancer Center, Kita-adachi-gun, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Toranomon Hospital, Minato, Tokyo
  - Akita University Hospital, Akita
  - Fukushima Medical University Hospital, Fukushima
  - Gifu University Hospital, Gifu
  - Hiroshima Prefectural Hospital, Hiroshima
  - Kyoto University Hospital, Kyoto
  - Okayama University Hospital, Okayama

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Bando H, Ueda A, Terata K, Doi M, Nagai SE, Hattori M, Watanabe K, Tamura N, Futamura M, Koizumi K, Niikura N, Miyaji T, Muramatsu Y, Xu L, Masuda N, Saji S. Health-related quality of life and physical activity collected via mobile application and wearable device in patients with HR +/HER2 - advanced breast cancer treated with palbociclib plus endocrine therapy or endocrine therapy alone: 6-month longitudinal study (JBCRG-26). Breast Cancer. 2025 Sep;32(5):1132-1143. doi: 10.1007/s12282-025-01744-0. Epub 2025 Jul 18. PMID 40681949
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, multicenter, observational study evaluated patient reported outcome (PRO) and physical activity using smartphone-based application and wearable device in Japanese participants diagnosed with hormone receptor positive (HR+) /human epidermal growth factor receptor 2 negative (HER2-) advanced breast cancer (ABC), who received palbociclib plus endocrine therapy or endocrine monotherapy.
Pre-assignment Details: A total of 99 participants were enrolled into the study and were observed for maximum up to 24 Weeks.
Groups:
- Group 1: Palbociclib Plus Endocrine Therapy: Participants with HR+/HER2- ABC who received palbociclib plus endocrine therapy based on the discretion of the treating physician under routine clinical practice were included. Palbociclib was administered for 3 consecutive weeks followed by 1 week off treatment to comprise one cycle of 4 weeks.
- Group 2: Endocrine Monotherapy: Participants with HR+/HER2- ABC who received endocrine monotherapy based on the discretion of the treating physician under routine clinical practice were included. One cycle was of 4 weeks.
Period: Overall Study
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Started | 78 | 21
Completed | 74 | 20
Not Completed | 4 | 1
Not completed — Progressive disease | 3 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Evaluable population included all eligible participants who were enrolled in the study and who responded to at least 1 item or measured at least 1 metrics of study application or device. Participants were analyzed according to the enrolled group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy | Total
Number analyzed (Participants) | 78 | 21 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.2 (10.0) | 56.3 (10.1) | 57.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 21 | 99
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 78 | 21 | 99
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-30 (Items) [EORTC-QLQ-C30] Global Health Status (GHS) Sub-scale Score for Cycle 1
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to evaluate cancer participants' quality of life (QOL), and it is composed of five multi-item functional subscales (physical, role, emotional, cognitive, and social functioning), three multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global health status scale (GHS)/QOL subscale, and six single item symptom scales assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and the financial impact of cancer). The GHS/QOL was scored on a 7-point Likert scale where 1=very much to 7=not at all. Responses to GHS/QOL subscales were converted to a 0 to 100 scale. For GHS/QOL subscale, higher scores indicated a better QOL. Baseline values were those measured between enrollment and the day before treatment start.
Time Frame: Baseline, Cycle 1 (1 cycle = 4 Weeks)
Population: Evaluable population included all eligible participants who were enrolled in the study and who responded to at least 1 item or measured at least 1 metrics of study application or device. Participants were analyzed according to the enrolled group. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 76 | 20
Units on a scale | 0.77 (19.25) | -0.42 (20.67)

2. Primary Outcome: Change From Baseline in EORTC-QLQ-C30 GHS Sub-scale Score for Cycle 2
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to evaluate cancer participants' QOL, and it is composed of five multi-item functional subscales (physical, role, emotional, cognitive, and social functioning), three multi-item symptom scales (fatigue, nausea/vomiting, and pain), a GHS/QOL subscale, and six single item symptom scales assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and the financial impact of cancer). The GHS/QOL was scored on a 7-point Likert scale where 1=very much to 7=not at all. Responses to GHS/QOL subscales were converted to a 0 to 100 scale. For GHS/QOL subscale, higher scores indicated a better QOL. Baseline values were those measured between enrollment and the day before treatment start.
Time Frame: Baseline, Cycle 2 (1 cycle = 4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 74 | 20
Units on a scale | 6.08 (21.38) | 0.42 (23.95)

3. Primary Outcome: Change From Baseline in EORTC-QLQ-C30 GHS Sub-scale Score for Cycle 3
Description: as for outcome 2
Time Frame: Baseline, Cycle 3 (1 cycle = 4 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 74 | 19
Units on a scale | 8.00 (21.61) | 5.70 (27.22)

4. Primary Outcome: Change From Baseline in EORTC-QLQ-C30 GHS Sub-scale Score for Cycle 4
Description: as for outcome 2
Time Frame: Baseline, Cycle 4 (1 cycle = 4 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 73 | 18
Units on a scale | 6.62 (20.50) | -0.93 (30.50)

5. Primary Outcome: Change From Baseline in EORTC-QLQ-C30 GHS Sub-scale Score for Cycle 5
Description: as for outcome 2
Time Frame: Baseline, Cycle 5 (1 cycle = 4 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 71 | 15
Units on a scale | 4.23 (20.79) | -2.78 (28.11)

6. Primary Outcome: Change From Baseline in EORTC-QLQ-C30 GHS Sub-scale Score for Cycle 6
Description: as for outcome 2
Time Frame: Baseline, Cycle 6 (1 cycle = 4 Weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 68 | 17
Units on a scale | 4.78 (22.78) | 2.94 (29.01)

7. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 1
Description: Sedentary time was used to assess physical activity metrics. Sedentary time was derived by Actigraph's algorithm based on raw data collected by Actigraph Insight Watch. Physical activity metrics were averaged at weekly basis which included 5 or more days of wearing the device for 10 hours or longer during a day except for bedtime.
Time Frame: Baseline, Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 75 | 21
Minutes | 18 (83) | 13 (100)

8. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 2
Description: as for outcome 7
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 74 | 20
Minutes | 8 (114) | -32 (130)

9. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 3
Description: as for outcome 7
Time Frame: Baseline, Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 72 | 19
Minutes | 12 (105) | -8 (159)

10. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 4
Description: as for outcome 7
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 70 | 18
Minutes | -5 (98) | -43 (173)

11. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 5
Description: as for outcome 7
Time Frame: Baseline, Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 73 | 18
Minutes | -7 (121) | -50 (149)

12. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 6
Description: as for outcome 7
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 67 | 17
Minutes | -13 (118) | -27 (146)

13. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 7
Description: as for outcome 7
Time Frame: Baseline, Week 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 72 | 16
Minutes | -9 (114) | -67 (186)

14. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 8
Description: as for outcome 7
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 71 | 15
Minutes | -5 (114) | -29 (125)

15. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 9
Description: as for outcome 7
Time Frame: Baseline, Week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 70 | 17
Minutes | -8 (130) | -20 (201)

16. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 10
Description: as for outcome 7
Time Frame: Baseline, Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 70 | 15
Minutes | -8 (130) | -4 (146)

17. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 11
Description: as for outcome 7
Time Frame: Baseline, Week 11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 67 | 17
Minutes | -16 (132) | -57 (207)

18. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 63 | 17
Minutes | -5 (137) | -66 (190)

19. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 13
Description: as for outcome 7
Time Frame: Baseline, Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 61 | 14
Minutes | -10 (145) | -14 (112)

20. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 14
Description: as for outcome 7
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 65 | 15
Minutes | -7 (138) | -14 (136)

21. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 15
Description: as for outcome 7
Time Frame: Baseline, Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 65 | 13
Minutes | -10 (134) | -60 (133)

22. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 16
Description: as for outcome 7
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 67 | 14
Minutes | -3 (128) | -45 (179)

23. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 17
Description: as for outcome 7
Time Frame: Baseline, Week 17
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 66 | 12
Minutes | -6 (128) | -18 (106)

24. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 18
Description: as for outcome 7
Time Frame: Baseline, Week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 64 | 13
Minutes | 2 (140) | -24 (134)

25. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 19
Description: as for outcome 7
Time Frame: Baseline, Week 19
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 62 | 12
Minutes | -2 (136) | -39 (82)

26. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 20
Description: as for outcome 7
Time Frame: Baseline, Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 61 | 11
Minutes | -6 (147) | -64 (179)

27. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 21
Description: as for outcome 7
Time Frame: Baseline, Week 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 61 | 13
Minutes | 11 (145) | -32 (178)

28. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 22
Description: as for outcome 7
Time Frame: Baseline, Week 22
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 62 | 15
Minutes | 2 (138) | -46 (143)

29. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 23
Description: as for outcome 7
Time Frame: Baseline, Week 23
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 62 | 12
Minutes | -1 (140) | -70 (128)

30. Primary Outcome: Change From Baseline in Sedentary Time Wearing at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 61 | 15
Minutes | -22 (161) | -102 (176)

31. Secondary Outcome: Change From Baseline in EORTC-QLQ-C30 Functional Sub-scale Scores at Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to evaluate cancer patients' QOL, and it's composed of five multi-item functional subscales (physical [P], role [R], emotional [E], cognitive [C], and social [S] functioning [F]). Response to functional scales is based on a 4-point Likert scale and ranges from 'not at all' to 'very much'. Responses to all functional sub-scales were converted to a 0 to 100 scale. For functional sub-scale, higher scores indicated a better level of functioning.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle=4 weeks)
Population: Evaluable population included all eligible participants who were enrolled in the study and who responded to at least 1 item or measured at least 1 metrics of study application or device. Participants were analyzed according to the enrolled group. All participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants analyzed for the specific timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 78 | 21
Units on a scale
  PF: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  PF: Change at Cycle 1 | -1.58 (14.6) | -2.33 (15.93)
  PF: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  PF: Change at Cycle 2 | 3.15 (14.14) | 1.33 (11.77)
  PF: Change at Cycle 3: number analyzed (Participants) | 74 | 19
  PF: Change at Cycle 3 | 1.53 (16.65) | 1.75 (14.2)
  PF: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  PF: Change at Cycle 4 | 3.11 (17.43) | -1.11 (10.29)
  PF: Change at Cycle5: number analyzed (Participants) | 71 | 15
  PF: Change at Cycle5 | 2.72 (19.7) | -8.44 (17.9)
  PF: Change at Cycle 6: number analyzed (Participants) | 68 | 17
  PF: Change at Cycle 6 | 0.39 (18.71) | -1.18 (13.99)
  RF: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  RF: Change at Cycle 1 | -1.75 (23.03) | -4.17 (16.11)
  RF: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  RF: Change at Cycle 2 | 2.03 (20.26) | -1.67 (20.16)
  RF Change at Cycle 3: number analyzed (Participants) | 74 | 19
  RF Change at Cycle 3 | 4.28 (21.02) | -4.39 (19.12)
  RF: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  RF: Change at Cycle 4 | 2.97 (22.8) | -4.63 (29.6)
  RF Change at Cycle 5: number analyzed (Participants) | 71 | 15
  RF Change at Cycle 5 | 2.35 (24.12) | -10 (23.4)
  RF Change at Cycle 6: number analyzed (Participants) | 68 | 17
  RF Change at Cycle 6 | 0.98 (25.58) | -2.94 (24.46)
  EF: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  EF: Change at Cycle 1 | 8.22 (16.69) | 0.83 (16.42)
  EF: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  EF: Change at Cycle 2 | 10.59 (18.21) | -2.5 (10.85)
  EF: Change at Cycle 3: number analyzed (Participants) | 74 | 19
  EF: Change at Cycle 3 | 10.36 (16.31) | -1.75 (12.9)
  EF: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  EF: Change at Cycle 4 | 9.25 (19.12) | -5.09 (19.83)
  EF: Change at Cycle 5: number analyzed (Participants) | 71 | 15
  EF: Change at Cycle 5 | 8.8 (18.57) | -2.22 (11.12)
  EF: Change at Cycle 6: number analyzed (Participants) | 68 | 17
  EF: Change at Cycle 6 | 9.31 (16.64) | -3.43 (15.33)
  CF: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  CF: Change at Cycle 1 | 1.75 (16.46) | -2.5 (19.7)
  CF: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  CF: Change at Cycle 2 | 1.13 (16.16) | -3.33 (17.61)
  CF: Change at Cycle 3: number analyzed (Participants) | 74 | 19
  CF: Change at Cycle 3 | 0.23 (16.44) | -7.02 (23.12)
  CF: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  CF: Change at Cycle 4 | -091 (20.39) | -8.33 (20.01)
  CF: Change at Cycle 5: number analyzed (Participants) | 71 | 15
  CF: Change at Cycle 5 | -2.58 (19.03) | -2.22 (22.6)
  CF: Change at Cycle 6: number analyzed (Participants) | 68 | 17
  CF: Change at Cycle 6 | -3.19 (21.01) | -7.84 (23.66)
  SF: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  SF: Change at Cycle 1 | 1.32 (21.39) | -0.83 (14.78)
  SF: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  SF: Change at Cycle 2 | 2.7 (22.25) | 4.17 (20.86)
  SF: Change at Cycle 3: number analyzed (Participants) | 74 | 19
  SF: Change at Cycle 3 | 1.35 (22.03) | 4.39 (19.12)
  SF: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  SF: Change at Cycle 4 | -0.68 (23.31) | -2.78 (18.3)
  SF: Change at Cycle 5: number analyzed (Participants) | 71 | 15
  SF: Change at Cycle 5 | -1.17 (24.29) | -6.67 (25.04)
  SF: Change at Cycle 6: number analyzed (Participants) | 68 | 17
  SF: Change at Cycle 6 | -2.45 (21.98) | 1.96 (18.52)

32. Secondary Outcome: Change From Baseline in EORTC-QLQ-C30 Symptomatic Sub-scale Scores at Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to evaluate cancer patients' QOL, and it's composed of three multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global QOL) subscale, and six single item symptom scales assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and the financial impact of cancer). Response to symptom sub-scales is based on a 4-point Likert scale and a higher score indicated more severe symptoms. Responses to all symptom sub-scales were converted to a 0 to 100 scale. A higher score indicated more severe symptoms. A 10-point or higher change in scores from baseline was considered clinically significant.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle=4 weeks)
Population: Evaluable population included all eligible participants who were enrolled in the study and who responded at least 1 item or measured at least 1 metrics of study application or device. Participants were analyzed according to the enrolled group. All participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specific timepoints.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 78 | 21
Units on a scale
  Fatigue: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  Fatigue: Change at Cycle 1 | 0.15 (17.54) | -1.11 (16.48)
  Fatigue: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  Fatigue: Change at Cycle 2 | -2.4 (16.27) | -0.56 (20.86)
  Fatigue: Change at Cycle 3: number analyzed (Participants) | 74 | 19
  Fatigue: Change at Cycle 3 | -3.3 (18.18) | -4.68 (19)
  Fatigue: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  Fatigue: Change at Cycle 4 | -1.52 (21.14) | 3.7 (21.56)
  Fatigue: Change at Cycle 5: number analyzed (Participants) | 71 | 15
  Fatigue: Change at Cycle 5 | -0.78 (22.72) | 3.7 (25.77)
  Fatigue: Change at Cycle 6: number analyzed (Participants) | 68 | 17
  Fatigue: Change at Cycle 6 | -0.49 (23.39) | -1.31 (18.79)
  Nausea, Vomiting: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  Nausea, Vomiting: Change at Cycle 1 | 0.66 (16.2) | -4.17 (25.86)
  Nausea, Vomiting: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  Nausea, Vomiting: Change at Cycle 2 | -2.03 (12.93) | -5.83 (23.12)
  Nausea, Vomiting: Change at Cycle 3: number analyzed (Participants) | 74 | 19
  Nausea, Vomiting: Change at Cycle 3 | -1.13 (15.44) | -6.14 (23.71)
  Nausea, Vomiting: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  Nausea, Vomiting: Change at Cycle 4 | -3.2 (14.61) | -7.41 (24.4)
  Nausea, Vomiting: Change at Cycle 5: number analyzed (Participants) | 71 | 15
  Nausea, Vomiting: Change at Cycle 5 | -2.58 (15.85) | -6.67 (28.73)
  Nausea, Vomiting: Change at Cycle 6: number analyzed (Participants) | 68 | 17
  Nausea, Vomiting: Change at Cycle 6 | -3.43 (13.37) | -5.88 (26.31)
  Pain: Change at Cycle 1: number analyzed (Participants) | 76 | 20
  Pain: Change at Cycle 1 | -0.88 (16.75) | 4.17 (16.99)
  Pain: Change at Cycle 2: number analyzed (Participants) | 74 | 20
  Pain: Change at Cycle 2 | -4.73 (19.99) | 1.67 (23.51)
  Pain: Change at Cycle 3: number analyzed (Participants) | 74 | 19
  Pain: Change at Cycle 3 | -5.86 (22.65) | -3.51 (24.58)
  Pain: Change at Cycle 4: number analyzed (Participants) | 73 | 18
  Pain: Change at Cycle 4 | -5.02 (26.01) | 2.78 (28.73)
  Pain: Change at Cycle 5: number analyzed (Participants) | 71 | 15
  Pain: Change at Cycle 5 | -5.4 (25.94) | 12.22 (24.77)
  Pain: Change at Cycle 6: number analyzed (Participants) | 68 | 17
  Pain: Change at Cycle 6 | 0 (24.43) | 2.94 (23)

33. Secondary Outcome: Change From Baseline in Steps Taken at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Description: Total estimated steps taken per week were reported in this outcome measure.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Steps per week
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 78 | 21
Steps per week
  Change at Week 1: number analyzed (Participants) | 75 | 21
  Change at Week 1 | -164 (927) | -340 (1219)
  Change at Week 2: number analyzed (Participants) | 74 | 20
  Change at Week 2 | 0 (996) | -39 (1413)
  Change at Week 3: number analyzed (Participants) | 72 | 19
  Change at Week 3 | -17 (1104) | -397 (1349)
  Change at Week 4: number analyzed (Participants) | 70 | 18
  Change at Week 4 | -17 (1004) | 13 (1608)
  Change at Week 5: number analyzed (Participants) | 73 | 18
  Change at Week 5 | 171 (1031) | 165 (1618)
  Change at Week 6: number analyzed (Participants) | 67 | 17
  Change at Week 6 | 353 (1253) | 54 (1468)
  Change at Week 7: number analyzed (Participants) | 72 | 16
  Change at Week 7 | 82 (1199) | -425 (1388)
  Change at Week 8: number analyzed (Participants) | 71 | 15
  Change at Week 8 | 147 (1376) | 481 (1733)
  Change at Week 9: number analyzed (Participants) | 70 | 17
  Change at Week 9 | 263 (1242) | -102 (1962)
  Change at Week 10: number analyzed (Participants) | 70 | 15
  Change at Week 10 | 279 (1470) | 251 (1869)
  Change at Week 11: number analyzed (Participants) | 67 | 17
  Change at Week 11 | 82 (1324) | 177 (1882)
  Change at Week 12: number analyzed (Participants) | 63 | 17
  Change at Week 12 | 260 (1514) | 168 (1806)
  Change at Week 13: number analyzed (Participants) | 61 | 14
  Change at Week 13 | 285 (1355) | 940 (1808)
  Change at Week 14: number analyzed (Participants) | 65 | 15
  Change at Week 14 | 395 (1526) | 389 (1787)
  Change at Week 15: number analyzed (Participants) | 65 | 13
  Change at Week 15 | 79 (1490) | 267 (1787)
  Change at Week 16: number analyzed (Participants) | 67 | 14
  Change at Week 16 | 188 (1540) | 387 (2142)
  Change at Week 17: number analyzed (Participants) | 66 | 12
  Change at Week 17 | 81 (1477) | 718 (1743)
  Change at Week 18: number analyzed (Participants) | 64 | 13
  Change at Week 18 | 207 (1418) | 264 (2274)
  Change at Week 19: number analyzed (Participants) | 62 | 12
  Change at Week 19 | 174 (1495) | 155 (2092)
  Change at Week 20: number analyzed (Participants) | 61 | 11
  Change at Week 20 | 254 (1234) | 726 (1820)
  Change at Week 21: number analyzed (Participants) | 61 | 13
  Change at Week 21 | 518 (1478) | 166 (2082)
  Change at Week 22: number analyzed (Participants) | 62 | 15
  Change at Week 22 | 334 (1174) | 362 (1875)
  Change at Week 23: number analyzed (Participants) | 62 | 12
  Change at Week 23 | 321 (1579) | 691 (1865)
  Change at Week 24: number analyzed (Participants) | 61 | 15
  Change at Week 24 | 447 (1860) | 202 (1690)

34. Secondary Outcome: Change From Baseline for Moderate to Vigorous Physical Activity (MVPA) Time at Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Description: Total estimated number of minutes of moderate or higher (moderate to vigorous) physical activity per date as calculated using the Staudenmayer '15 technique were reported in this outcome measure.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: Evaluable population included all eligible participants who were enrolled in the study and who responded to at least 1 item or measured at least 1 metrics of study application or device. Participants were analyzed according to the enrolled group. All participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specific timepoints.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 78 | 21
Minutes
  Change at Week 1: number analyzed (Participants) | 75 | 21
  Change at Week 1 | -1 (28) | -7 (20)
  Change at Week 2: number analyzed (Participants) | 74 | 20
  Change at Week 2 | -1 (38) | -9 (20)
  Change at Week 3: number analyzed (Participants) | 72 | 19
  Change at Week 3 | -4 (32) | -10 (22)
  Change at Week 4: number analyzed (Participants) | 70 | 18
  Change at Week 4 | -2 (41) | -2 (27)
  Change at Week 5: number analyzed (Participants) | 73 | 18
  Change at Week 5 | 5 (48) | -4 (23)
  Change at Week 6: number analyzed (Participants) | 67 | 17
  Change at Week 6 | 4 (35) | -5 (27)
  Change at Week 7: number analyzed (Participants) | 72 | 16
  Change at Week 7 | -3 (58) | -12 (24)
  Change at Week 8: number analyzed (Participants) | 71 | 15
  Change at Week 8 | -2 (49) | 1 (16)
  Change at Week 9: number analyzed (Participants) | 70 | 17
  Change at Week 9 | 5 (55) | -6 (26)
  Change at Week 10: number analyzed (Participants) | 70 | 15
  Change at Week 10 | -1 (57) | 0 (23)
  Change at Week 11: number analyzed (Participants) | 67 | 17
  Change at Week 11 | -2 (47) | -4 (28)
  Change at Week 12: number analyzed (Participants) | 63 | 17
  Change at Week 12 | 1 (50) | -6 (19)
  Change at Week 13: number analyzed (Participants) | 61 | 14
  Change at Week 13 | 2 (51) | 10 (21)
  Change at Week 14: number analyzed (Participants) | 65 | 15
  Change at Week 14 | 1 (58) | 1 (22)
  Change at Week 15: number analyzed (Participants) | 65 | 13
  Change at Week 15 | 0 (68) | -2 (20)
  Change at Week 16: number analyzed (Participants) | 67 | 14
  Change at Week 16 | -2 (55) | -8 (29)
  Change at Week 17: number analyzed (Participants) | 66 | 12
  Change at Week 17 | -6 (47) | 0 (24)
  Change at Week 18: number analyzed (Participants) | 64 | 13
  Change at Week 18 | -5 (59) | 1 (26)
  Change at Week 19: number analyzed (Participants) | 62 | 12
  Change at Week 19 | -5 (64) | -9 (36)
  Change at Week 20: number analyzed (Participants) | 61 | 11
  Change at Week 20 | -6 (44) | 0 (30)
  Change at Week 21: number analyzed (Participants) | 61 | 13
  Change at Week 21 | -1 (51) | -11 (25)
  Change at Week 22: number analyzed (Participants) | 62 | 15
  Change at Week 22 | -2 (40) | -5 (32)
  Change at Week 23: number analyzed (Participants) | 62 | 12
  Change at Week 23 | 3 (53) | 3 (33)
  Change at Week 24: number analyzed (Participants) | 61 | 15
  Change at Week 24 | 3 (49) | -4 (23)

35. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Grade 3 or Higher AEs and Treatment Related Adverse Events
Description: AE= any untoward medical occurrence,could therefore be any unfavorable,unintended sign (including an abnormal laboratory finding),symptom,or disease,whether or not related to the participant's participation in the study. An SAE was any untoward medical occurrence at any dose that:resulted in death;was life-threatening(LT);required inpatient hospitalization or prolongation of existing hospitalization;resulted in persistent or significant disability/incapacity(substantial disruption of the ability to conduct normal life functions);resulted in congenital anomaly/birth defect;or an important medical event. AEs were graded(G) according to Common Terminology Criteria for AE(CTCAE) version 4.03. G3 (Severe AE),G4 (LT consequences;urgent intervention indicated),G5 (Death related to AE). TEAEs were those events with onset dates occurring during the on-treatment period (the time from start of study treatment up to 28 days after last dose). Relatedness was based on the investigator's judgement.
Time Frame: From start of study treatment up to 28 days after last dose of treatment (Up to 28 weeks)
Population: Safety Analysis set included all participants who received at least 1 dose of palbociclib or endocrine therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 78 | 21
Participants
  Adverse Events | 68 | 5
  Serious Adverse Events | 3 | 0
  Grade 3 or Higher AEs | 54 | 1
  Treatment Related Adverse Events | 66 | 5

36. Secondary Outcome: Number of Participants According to Fatigue Severity Based on Patient Reported Outcome - Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a PRO measurement system that includes a library of questions that measures symptomatic adverse events from the participant perspective. Participants were required to provide their responses to the questions on fatigue severity on a five-point Likert scale. For Fatigue Severity (FS) scoring was as follows: 0= None, 10= Mild, 20= Moderate, 30= Severe, 40= Very Severe.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle=4 weeks)
Population: Evaluable population included all eligible participants who were enrolled in the study and who responded to at least 1 item or measured at least 1 metrics of study application or device. Participants were analyzed according to the enrolled group. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies number of participants evaluable for the specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 77 | 21
Participants
  FS: Baseline: None | 27 | 5
  FS: Baseline: Mild | 32 | 10
  FS: Baseline: Moderate | 11 | 4
  FS: Baseline: Severe | 7 | 2
  FS: Baseline: Very Severe | 0 | 0
  FS: Cycle 1: None | 4 | 4
  FS: Cycle 1: Mild | 35 | 8
  FS: Cycle 1: Moderate | 27 | 6
  FS: Cycle 1: Severe | 9 | 3
  FS: Cycle 1: Very Severe | 2 | 0
  FS: Cycle 2: number analyzed (Participants) | 76 | 20
  FS: Cycle 2: None | 6 | 4
  FS: Cycle 2: Mild | 41 | 7
  FS: Cycle 2: Moderate | 20 | 7
  FS: Cycle 2: Severe | 7 | 1
  FS: Cycle 2: Very Severe | 2 | 1
  FS: Cycle 3: number analyzed (Participants) | 75 | 21
  FS: Cycle 3: None | 10 | 5
  FS: Cycle 3: Mild | 40 | 8
  FS: Cycle 3: Moderate | 17 | 6
  FS: Cycle 3: Severe | 8 | 1
  FS: Cycle 3: Very Severe | 0 | 1
  FS: Cycle 4: number analyzed (Participants) | 75 | 19
  FS: Cycle 4: None | 8 | 3
  FS: Cycle 4: Mild | 41 | 6
  FS: Cycle 4: Moderate | 19 | 9
  FS: Cycle 4: Severe | 6 | 1
  FS: Cycle 4: Very Severe | 1 | 0
  FS: Cycle 5: number analyzed (Participants) | 72 | 17
  FS: Cycle 5: None | 8 | 3
  FS: Cycle 5: Mild | 38 | 6
  FS: Cycle 5: Moderate | 20 | 5
  FS: Cycle 5: Severe | 6 | 3
  FS: Cycle 5: Very Severe | 0 | 0
  FS: Cycle 6: number analyzed (Participants) | 68 | 17
  FS: Cycle 6: None | 9 | 3
  FS: Cycle 6: Mild | 34 | 8
  FS: Cycle 6: Moderate | 14 | 4
  FS: Cycle 6: Severe | 9 | 1
  FS: Cycle 6: Very Severe | 2 | 1

37. Secondary Outcome: Number of Participants According to Fatigue Interference Based on PRO-CTCAE
Description: The PRO-CTCAE is a PRO measurement system that includes a library of questions that measures symptomatic adverse events from the participant perspective. Participants were required to provide their responses to the questions on fatigue interference on a five-point Likert scale. For Fatigue Interference (FI) scoring was as follows: 0= Not at all/None/Never, 1= A Little bit, 2: Somewhat, 3= Quite a bit, 4= Very much.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle=4 weeks)
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 77 | 21
Participants
  FI: Baseline: Not at all/None/Never | 33 | 6
  FI: Baseline: A Little bit | 30 | 10
  FI: Baseline: Somewhat | 8 | 2
  FI: Baseline: Quite a bit | 3 | 2
  FI: Baseline: Very Much | 3 | 1
  FI: Cycle 1: Not at all/None/Never | 14 | 7
  FI: Cycle 1: A Little bit | 32 | 8
  FI: Cycle 1: Somewhat | 23 | 4
  FI: Cycle 1: Quite a bit | 6 | 2
  FI: Cycle 1: Very Much | 2 | 0
  FI: Cycle 2: number analyzed (Participants) | 76 | 20
  FI: Cycle 2: Not at all/None/Never | 13 | 4
  FI: Cycle 2: A Little bit | 42 | 9
  FI: Cycle 2: Somewhat | 13 | 5
  FI: Cycle 2: Quite a bit | 7 | 1
  FI: Cycle 2: Very Much | 1 | 1
  FI: Cycle 3: number analyzed (Participants) | 75 | 21
  FI: Cycle 3: Not at all/None/Never | 19 | 7
  FI: Cycle 3: A Little bit | 36 | 8
  FI: Cycle 3: Somewhat | 13 | 4
  FI: Cycle 3: Quite a bit | 6 | 0
  FI: Cycle 3: Very Much | 1 | 2
  FI: Cycle 4: number analyzed (Participants) | 75 | 19
  FI: Cycle 4: Not at all/None/Never | 19 | 3
  FI: Cycle 4: A Little bit | 32 | 8
  FI: Cycle 4: Somewhat | 17 | 6
  FI: Cycle 4: Quite a bit | 5 | 2
  FI: Cycle 4: Very Much | 2 | 0
  FI: Cycle 5: number analyzed (Participants) | 72 | 17
  FI: Cycle 5: Not at all/None/Never | 17 | 4
  FI: Cycle 5: A Little bit | 32 | 7
  FI: Cycle 5: Somewhat | 15 | 4
  FI: Cycle 5: Quite a bit | 7 | 2
  FI: Cycle 5: Very Much | 1 | 0
  FI: Cycle 6: number analyzed (Participants) | 68 | 17
  FI: Cycle 6: Not at all/None/Never | 18 | 4
  FI: Cycle 6: A Little bit | 29 | 8
  FI: Cycle 6: Somewhat | 12 | 2
  FI: Cycle 6: Quite a bit | 7 | 2
  FI: Cycle 6: Very Much | 2 | 1

38. Secondary Outcome: Number of Participants According to Pain Severity Based on PRO-CTCAE
Description: The PRO-CTCAE is a PRO measurement system that includes a library of questions that measures symptomatic adverse events from the participant perspective. Participants were required to provide their responses to the questions on pain severity on a five-point Likert scale. For Pain Severity (PS) scoring was as follows: 0= None, 10= Mild, 20= Moderate, 30= Severe, 40= Very Severe.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle=4 weeks)
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 77 | 21
Participants
  PS: Baseline: None | 22 | 10
  PS: Baseline: Mild | 33 | 6
  PS: Baseline: Moderate | 16 | 4
  PS: Baseline: Severe | 4 | 1
  PS: Baseline: Very Severe | 2 | 0
  PS: Cycle 1: None | 8 | 6
  PS: Cycle 1: Mild | 31 | 7
  PS: Cycle 1: Moderate | 27 | 5
  PS: Cycle 1: Severe | 9 | 3
  PS: Cycle 1: Very Severe | 2 | 0
  PS: Cycle 2: number analyzed (Participants) | 76 | 20
  PS: Cycle 2: None | 12 | 3
  PS: Cycle 2: Mild | 43 | 8
  PS: Cycle 2: Moderate | 15 | 8
  PS: Cycle 2: Severe | 5 | 0
  PS: Cycle 2: Very Severe | 1 | 1
  PS: Cycle 3: number analyzed (Participants) | 75 | 21
  PS: Cycle 3: None | 15 | 4
  PS: Cycle 3: Mild | 37 | 10
  PS: Cycle 3: Moderate | 14 | 5
  PS: Cycle 3: Severe | 9 | 2
  PS: Cycle 3: Very Severe | 0 | 0
  PS: Cycle 4: number analyzed (Participants) | 75 | 19
  PS: Cycle 4: None | 16 | 2
  PS: Cycle 4: Mild | 35 | 12
  PS: Cycle 4: Moderate | 18 | 4
  PS: Cycle 4: Severe | 4 | 1
  PS: Cycle 4: Very Severe | 2 | 0
  PS: Cycle 5: number analyzed (Participants) | 72 | 17
  PS: Cycle 5: None | 15 | 3
  PS: Cycle 5: Mild | 35 | 6
  PS: Cycle 5: Moderate | 15 | 4
  PS: Cycle 5: Severe | 6 | 4
  PS: Cycle 5: Very Severe | 1 | 0
  PS: Cycle 6: number analyzed (Participants) | 68 | 17
  PS: Cycle 6: None | 14 | 3
  PS: Cycle 6: Mild | 30 | 7
  PS: Cycle 6: Moderate | 14 | 5
  PS: Cycle 6: Severe | 8 | 2
  PS: Cycle 6: Very Severe | 2 | 0

39. Secondary Outcome: Number of Participants According to Pain Interference Based on PRO-CTCAE
Description: The PRO-CTCAE is a PRO measurement system that includes a library of questions that measures symptomatic adverse events from the participant perspective. Participants were required to provide their responses to the questions on pain interference on a five-point Likert scale. For Pain Interference (PI) scoring was as follows: 0= Not at all/None/Never, 1= A Little bit, 2: Somewhat, 3= Quite a bit, 4= Very much.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle=4 weeks)
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 77 | 21
Participants
  PI: Baseline: Not at all/None/Never | 39 | 12
  PI: Baseline: A Little bit | 24 | 6
  PI: Baseline: Somewhat | 8 | 2
  PI: Baseline: Quite a bit | 4 | 0
  PI: Baseline: Very Much | 2 | 1
  PI: Cycle 1: Not at all/None/Never | 20 | 8
  PI: Cycle 1: A Little bit | 28 | 8
  PI: Cycle 1: Somewhat | 18 | 3
  PI: Cycle 1: Quite a bit | 8 | 2
  PI: Cycle 1: Very Much | 3 | 0
  PI: Cycle 2: number analyzed (Participants) | 76 | 20
  PI: Cycle 2: Not at all/None/Never | 24 | 6
  PI: Cycle 2: A Little bit | 36 | 9
  PI: Cycle 2: Somewhat | 10 | 4
  PI: Cycle 2: Quite a bit | 3 | 1
  PI: Cycle 2: Very Much | 3 | 0
  PI: Cycle 3: number analyzed (Participants) | 75 | 21
  PI: Cycle 3: Not at all/None/Never | 26 | 8
  PI: Cycle 3: A Little bit | 32 | 7
  PI: Cycle 3: Somewhat | 11 | 5
  PI: Cycle 3: Quite a bit | 5 | 1
  PI: Cycle 3: Very Much | 1 | 0
  PI: Cycle 4: number analyzed (Participants) | 75 | 19
  PI: Cycle 4: Not at all/None/Never | 29 | 6
  PI: Cycle 4: A Little bit | 23 | 7
  PI: Cycle 4: Somewhat | 17 | 5
  PI: Cycle 4: Quite a bit | 4 | 1
  PI: Cycle 4: Very Much | 2 | 0
  PI: Cycle 5: number analyzed (Participants) | 72 | 17
  PI: Cycle 5: Not at all/None/Never | 26 | 4
  PI: Cycle 5: A Little bit | 25 | 6
  PI: Cycle 5: Somewhat | 14 | 3
  PI: Cycle 5: Quite a bit | 6 | 4
  PI: Cycle 5: Very Much | 1 | 0
  PI: Cycle 6: number analyzed (Participants) | 68 | 17
  PI: Cycle 6: Not at all/None/Never | 23 | 4
  PI: Cycle 6: A Little bit | 27 | 8
  PI: Cycle 6: Somewhat | 7 | 4
  PI: Cycle 6: Quite a bit | 9 | 1
  PI: Cycle 6: Very Much | 2 | 0

40. Secondary Outcome: Number of Participants According to Pain Frequency Based on PRO-CTCAE
Description: The PRO-CTCAE is a PRO measurement system that includes a library of questions that measures symptomatic adverse events from the participant perspective. Participants were required to provide their responses to the questions on pain frequency on a five-point Likert scale. For Pain Frequency (PF) scoring was as follows: 0= None, 1= Rarely, 2: Occasionally, 3= Frequently, 4=Almost Constantly.
Time Frame: Baseline, Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle=4 weeks)
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 77 | 21
Participants
  PF: Baseline: None | 18 | 8
  PF: Baseline: Rarely | 14 | 4
  PF: Baseline: Occasionally | 34 | 6
  PF: Baseline: Frequently | 7 | 1
  PF: Baseline: Almost Constantly | 4 | 2
  PF: Cycle 1: None | 7 | 4
  PF: Cycle 1: Rarely | 12 | 5
  PF: Cycle 1: Occasionally | 39 | 7
  PF: Cycle 1: Frequently | 9 | 4
  PF: Cycle 1: Almost Constantly | 10 | 1
  PF: Cycle 2: number analyzed (Participants) | 76 | 20
  PF: Cycle 2: None | 11 | 3
  PF: Cycle 2: Rarely | 14 | 7
  PF: Cycle 2: Occasionally | 41 | 7
  PF: Cycle 2: Frequently | 5 | 1
  PF: Cycle 2: Almost Constantly | 5 | 2
  PF: Cycle 3: number analyzed (Participants) | 75 | 21
  PF: Cycle 3: None | 13 | 4
  PF: Cycle 3: Rarely | 20 | 6
  PF: Cycle 3: Occasionally | 28 | 8
  PF: Cycle 3: Frequently | 10 | 2
  PF: Cycle 3: Almost Constantly | 4 | 1
  PF: Cycle 4: number analyzed (Participants) | 75 | 19
  PF: Cycle 4: None | 15 | 2
  PF: Cycle 4: Rarely | 17 | 5
  PF: Cycle 4: Occasionally | 25 | 10
  PF: Cycle 4: Frequently | 13 | 2
  PF: Cycle 4: Almost Constantly | 5 | 0
  PF: Cycle 5: number analyzed (Participants) | 72 | 17
  PF: Cycle 5: None | 15 | 2
  PF: Cycle 5: Rarely | 13 | 3
  PF: Cycle 5: Occasionally | 23 | 7
  PF: Cycle 5: Frequently | 14 | 5
  PF: Cycle 5: Almost Constantly | 7 | 0
  PF: Cycle 6: number analyzed (Participants) | 68 | 17
  PF: Cycle 6: None | 10 | 2
  PF: Cycle 6: Rarely | 19 | 4
  PF: Cycle 6: Occasionally | 18 | 6
  PF: Cycle 6: Frequently | 14 | 5
  PF: Cycle 6: Almost Constantly | 7 | 0

41. Secondary Outcome: Sedentary Time Before and After Disease Progression: Group 1 and 2 Pooled
Description: Sedentary time was used to assess physical activity metrics. Sedentary time was derived by Actigraph's algorithm based on raw data collected by Actigraph Insight Watch. Physical activity metrics were averaged at weekly basis which included 5 or more days of wearing the device 10 hours or longer during a day except for bedtime. Disease progression was defined as greater than (>) 25% increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: Before and after disease progression during the observation period (maximum up to 24 weeks)
Population: Safety Analysis set included all participants who received at least 1 dose of palbociclib or endocrine therapy. As per statistical analysis plan, when associations for group 1 and 2 were similar, the data for group 1 and 2 were pooled. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Group 1 and Group 2 Pooled: Participants with HR+/HER2- ABC who received palbociclib plus endocrine therapy or endocrine monotherapy based on the discretion of the treating physician under routine clinical practice were included.
Arm/Group | Group 1 and Group 2 Pooled
Number analyzed (Participants) | 11
Minutes
  Before disease progression | 574 (246)
  After disease progression | 594 (266)

42. Secondary Outcome: Steps Taken Before and After Disease Progression: Group 1 and 2 Pooled
Description: Total estimated steps taken per week were reported in this outcome measure. Disease progression was defined as >25% increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: Before and after disease progression during the observation period (maximum up to 24 weeks)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: Steps per week
Arm/Group | Group 1 and Group 2 Pooled
Number analyzed (Participants) | 11
Steps per week
  Before disease progression | 3601 (1993)
  After disease progression | 3599 (2017)

43. Secondary Outcome: MVPA Before and After Disease Progression: Group 1 and 2 Pooled
Description: Total estimated number of minutes of Moderate or higher (moderate to vigorous) physical activity per date as calculated using the Staudenmayer '15 technique were reported in this outcome measure. Disease progression was defined as >25% increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: Before and after disease progression during the observation period (maximum up to 24 weeks)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 and Group 2 Pooled
Number analyzed (Participants) | 11
Minutes
  Before disease progression | 73 (25)
  After disease progression | 75 (30)

44. Secondary Outcome: EORTC-QLQ-C30 GHS and Functional Sub-scale Score Before and After Disease Progression: Group 1 and 2 Pooled
Description: The EORTC-QLQ-C30 is a 30-item questionnaire to evaluate cancer participants' QOL,it's composed of five multi-item functional subscales (physical [P],role [R],emotional [E],cognitive [C], and social [S] functioning [F], three multi-item symptom scales (fatigue,nausea/vomiting,pain) a GHS/QOL subscale,and six single item symptom scales assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation,diarrhea,and the financial impact of cancer). The GHS/QOL was scored on a 7-point Likert scale where 1=very much to 7=not at all. Response to functional scales is based on a 4-point Likert scale and ranges from 'not at all' to 'very much'. Responses to GHS/QOL and all functional sub-scales were converted to a 0 to 100 scale. For GHS/QOL and functional subscale, higher scores indicated a better QOL and better level of functioning, respectively. Disease progression was defined as >25% increase in sum of longest diameter of target lesions compared to baseline.
Time Frame: Before and after disease progression during the observation period (maximum up to 24 weeks)
Population: Safety Analysis set included all participants who received at least 1 dose of palbociclib or endocrine therapy. As per statistical analysis plan, when associations for group 1 and 2 were similar, the data for group 1 and 2 were pooled. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies number of participants evaluable for the specific rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1 and Group 2 Pooled
Number analyzed (Participants) | 12
Units on a scale
  GHS (Before disease progression) | 69.4 (17.5)
  GHS (After disease progression): number analyzed (Participants) | 10
  GHS (After disease progression) | 53.3 (30.0)
  Physical Functioning (Before disease progression) | 80.6 (15.2)
  Physical Functioning (After disease progression): number analyzed (Participants) | 10
  Physical Functioning (After disease progression) | 68.0 (30.1)
  Role Functioning (Before disease progression) | 86.1 (17.2)
  Role Functioning (After disease progression): number analyzed (Participants) | 10
  Role Functioning (After disease progression) | 65.0 (38.0)
  Social Functioning (Before disease progression) | 88.9 (16.4)
  Social Functioning (After disease progression): number analyzed (Participants) | 10
  Social Functioning (After disease progression) | 76.7 (27.4)

45. Secondary Outcome: Number of Participants With Treatment Satisfaction
Description: Treatment satisfaction was evaluated with single item question (eg,"How satisfied are you with your current breast cancer treatment?") using the smart phone application. Responses were provided on a four-point Likert scale (dissatisfied, neutral, satisfied, very satisfied).
Time Frame: Day 15 of Cycle 1, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6 (each cycle = 4 weeks)
Population: Safety Analysis set included all participants who received at least 1 dose of palbociclib or endocrine therapy. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies number of participants evaluable for the specific timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
Number analyzed (Participants) | 77 | 21
Participants
  Cycle 1: number analyzed (Participants) | 77 | 20
  Cycle 1: Dissatisfied | 1 | 1
  Cycle 1: Neutral | 40 | 10
  Cycle 1: Satisfied | 27 | 5
  Cycle 1: Very Satisfied | 9 | 4
  Cycle 2: number analyzed (Participants) | 75 | 20
  Cycle 2: Dissatisfied | 1 | 0
  Cycle 2: Neutral | 35 | 10
  Cycle 2: Satisfied | 29 | 7
  Cycle 2: Very Satisfied | 10 | 3
  Cycle 3: number analyzed (Participants) | 77 | 18
  Cycle 3: Dissatisfied | 1 | 0
  Cycle 3: Neutral | 33 | 7
  Cycle 3: Satisfied | 32 | 9
  Cycle 3: Very Satisfied | 11 | 2
  Cycle 4: number analyzed (Participants) | 75 | 20
  Cycle 4: Dissatisfied | 0 | 0
  Cycle 4: Neutral | 31 | 10
  Cycle 4: Satisfied | 33 | 7
  Cycle 4: Very Satisfied | 11 | 3
  Cycle 5: number analyzed (Participants) | 75 | 18
  Cycle 5: Dissatisfied | 1 | 0
  Cycle 5: Neutral | 30 | 5
  Cycle 5: Satisfied | 31 | 11
  Cycle 5: Very Satisfied | 13 | 2
  Cycle 6: number analyzed (Participants) | 73 | 20
  Cycle 6: Dissatisfied | 1 | 0
  Cycle 6: Neutral | 29 | 7
  Cycle 6: Satisfied | 34 | 11
  Cycle 6: Very Satisfied | 9 | 2

46. Secondary Outcome: Number of Participants According to Starting Dose of Palbociclib Treatment
Description: Number of participants according to starting dose of palbociclib treatment (125 milligrams [mg], 100 mg and 75 mg) is reported in this outcome measure. Baseline values are those measured between enrollment and the day before treatment start.
Time Frame: Baseline
Population: Safety Analysis set included all participants who received at least 1 dose of palbociclib or endocrine therapy. No participant received palbociclib treatment in Group 2. Hence, no data was reported for Group 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy
Number analyzed (Participants) | 78
Participants
  125 mg | 73
  100 mg | 5
  75 mg | 0

47. Secondary Outcome: Number of Participants Who Had Any Palbociclib Dose Reduction
Time Frame: Up to 24 Weeks
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy
Number analyzed (Participants) | 78
Participants | 44

48. Secondary Outcome: Number of Participants Who Had Any Palbociclib Dose Interruption
Time Frame: Up to 24 Weeks
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy
Number analyzed (Participants) | 78
Participants | 31

49. Secondary Outcome: Number of Participants With Cycle Delay in Palbociclib Treatment
Time Frame: Up to 24 Weeks
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy
Number analyzed (Participants) | 78
Participants | 58

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 28 days after last dose of study treatment (up to 28 weeks)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Group 1: Palbociclib Plus Endocrine Therapy | Group 2: Endocrine Monotherapy
All-Cause Mortality (participants affected / at risk) | 1/78 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/78 | 0/21
Other Adverse Events (participants affected / at risk) | 65/78 | 5/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Palbociclib Plus Endocrine Therapy (N=78) | Group 2: Endocrine Monotherapy (N=21)
Pneumonia bacterial (Infections and infestations) | 1 | 0
Death (General disorders) | 1 | 0
SARS-CoV-2 (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Palbociclib Plus Endocrine Therapy (N=78) | Group 2: Endocrine Monotherapy (N=21)
Anaemia (Blood and lymphatic system disorders) | 11 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 11 | 0
Neutropenia (Blood and lymphatic system disorders) | 41 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 11 | 0
Fatigue (General disorders) | 3 | 0
Malaise (General disorders) | 4 | 2
Oedema peripheral (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 14 | 0
Platelet count decreased (Investigations) | 4 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT04736576/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT04736576/SAP_001.pdf